CLINICAL TRIAL: NCT01857947
Title: Usefulness of Pro-adrenomedullin (MR proADM)as a Predictor of Outcome in Acute Exacerbations of COPD Visiting the Emergency Room
Brief Title: Prognosis Value of Pro-adrenomedullin in Acute Exacerbations of COPD in ER
Acronym: UTAPE BPCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ThermoFisher Scientific Brahms Biomarkers France (Industry)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: UTAPE01
Record Dates: First submitted 2013-05-16; First posted 2013-05-20 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Pulmonary Disease, Chronic Obstructive Patients Admitted in Emergency Department for Acute Exacerbation
Keywords: AECOPD Mr ProADM Biomarkers ER Outcome
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- AECOPD Mr proADM (No Intervention): Patients involved in this study will have a simple blood sample collected for Mr proADM assessment at the end of study
  Interventions: Other: AECOPD Mr proADM

INTERVENTIONS:
Other: AECOPD Mr proADM

SUMMARY:
The purpose of this study is to determine whether pro-adrenomedullin (Mr proADM)in addition to clinical evaluation is effective to predict outcome of acute exacerbations of COPD patients visiting the emergency room(ER).

DETAILED DESCRIPTION:
Acute exacerbation of COPD (AECOPD)are usual and frequent cause of admission in emergency room (ER). No validated clinical or biological predictor of evolution are available.

The main objective is to determine the prognosis value of Mr proADM in addition to the clinical risk stratification for AE COPD patients in ER.

Patients presenting with a AECOPD diagnosis in ER will have a blood sample collected and freezed at their admission. Mr proADM will be assessed at the end of the study. Clinicians in charge of patients will not have the result during the management of their patients. This study implies no change in the patients' management.

Data related to the patients'demographic,current exacerbation and basic COPD characteristics will be collected.

ELIGIBILITY:
Inclusion Criteria:

* patients > 40 years old
* Acute exacerbation of COPD

Exclusion Criteria:

* Medico social conditions not allowing home discharge
* Other causes of Dyspnea: Pneumothorax, pulmonary embolism, pulmonary oedema, lung cancer
* Pneumonia on chest ray
* acute respiratory distress requiring immediate ICU transfer

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Actual)
Dates: Start 2013-03; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
composite outcome measure | at Day 30
  Death, subsequently transfer to ICU, relapse, need to be ventilated after 24 hours of their admission in ER

SECONDARY OUTCOMES:
composite outcome | at Day 7 of ER admission
  Death, subsequently transfer to ICU, relapse, need to be ventilated after 24 hours of their admission in ER
correlation between Mr proADM and patients Severity | at Day 7 and Day 30 of ED admission
  Correlation between MR proADM and patient's severity

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Roche, MD PHD, Study Chair — Hotel Dieu Hospital Paris; Martin Dres, MD, Study Director — Hopital Bicêtre Le Krémlin Bicêtre; Pierre Hausfater, MD PHD, Principal Investigator — Pitié Salpétrière Hospital Paris
Locations (2):
- France (2):
  - Hôpital Lariboisière, Paris, Paris
  - Pitié Salpétrière Hospital, Paris, Paris